CLINICAL TRIAL: NCT05584618
Title: Evaluation of Antenatal Education on Fear of ChildBirth, Depression, Anxiety, Maternal Self-Efficacy, and Delivery Mode in Primiparous Pregnant Women: A Prospective Randomized Controlled Study
Brief Title: Effect of Antenatal Education on Fear of ChildBirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08.06.2022-73
Record Dates: First submitted 2022-10-01; First posted 2022-10-18 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Fear of Childbirth; Stress
Keywords: antenatal education; fear of childbirth; depression, anxiety; stress; maternal self-efficacy; mode of delivery
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): The women allocated in experimental group will be given antenatal education for 6 weeks
  Interventions: Other: Education
- control (No Intervention): The women allocated for the control group will receive prenatal care services routinely provided at the outpatient clinics of the same hospital

INTERVENTIONS:
Other: Education — education
  Arms: intervention

SUMMARY:
The aim of this study was to investigate the effects of antenatal education on birth fear, depression, anxiety, stress, maternal self-efficacy, and mode of delivery in primiparous pregnant women

DETAILED DESCRIPTION:
There is still a lack of evidence regarding the effects of antenatal education on birth fear, maternal self-efficacy, anxiety, stress, depression, and mode of delivery. Therefore, this study aimed to investigate the effects of antenatal education on birth fear, anxiety, stress, depression, maternal self-efficacy, and mode of delivery

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Childbirth at fullterm (born at 38-42 weeks)
* Nulliparous women
* Women between the ages of 18-35
* Singleton pregnancy in 20 and 36 weeks of gestation
* Having a healthy newborn
* No participation in another prenatal program
* Absence of any psychiatric illness or comorbidities
* No use medications for a diagnosed mental disorder
* Baby with normal birth weight and APGAR score of 8 and above
* Women who have not developed postpartum complications
* Women without complicated/high-risk pregnancies, who do not experience a perinatal death or stillbirth
* Speaks and understands Turkish
* Women with a total fear of childbirth score W-DEQ-A ≥60 will be included.
* Women who give birth through vaginal route

Exclusion Criteria:

• Women who do not meet the sample selection criteria

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | at 20 to 36 weeks gestational age
  The scale developed by Cohen, Kamarck and Mermelstein (1983) and its Turkish adaptation was carried out by Eskin, Harlak, Demirkıran and Dereboy (2013), which aims to measure how stressful some situations in a person's life are perceived, consists of 14 items. The "Perceived Stress Scale" consists of the dimensions of "Perception of Inadequate Self-Efficacy" and "Perception of Stress/Discomfort". Participants evaluated each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". The internal consistency coefficient of the Turkish scale was 0.84 and the test-retest reliability was 0.87.
Perceived Stress Scale (PSS) | 6-8 weeks postpartum
  The scale developed by Cohen, Kamarck and Mermelstein (1983) and its Turkish adaptation was carried out by Eskin, Harlak, Demirkıran and Dereboy (2013), which aims to measure how stressful some situations in a person's life are perceived, consists of 14 items. The "Perceived Stress Scale" consists of the dimensions of "Perception of Inadequate Self-Efficacy" and "Perception of Stress/Discomfort". Participants evaluated each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". The internal consistency coefficient of the Turkish scale was 0.84 and the test-retest reliability was 0.87.
Wijma Delivery Expectancy/ Experience Questionnaire (W-DEQ- A) | at 20 to 36 weeks gestational age
  The scale was developed by Klaas and Barbro Wijma to measure the fear of childbirth and its Turkish adaptation and validity and reliability were conducted by Körükçü, Kukulu, and Fırat (2012, 2018). The scale consists of 33 items and the answers are enumerated between 0 and 5 as a 6-item liker scale, in which 0 means "completely" and 5 means "none". The range of the total score of the scale is between 0 and 165. The higher the scores, the higher the fear of birth experienced by women
Multidimensional Scale of Perceived Social Support (MSPSS) | at 20 to 36 weeks gestational age
  The scale developed by Zimet et al. in 1988 and Turkish adaptation, validity and reliability studies were carried out by Eker, Arkar, and Yaldız (2001). The MSPSS is a 12-item scale, and includes 3 groups about the source of support, each of which consisting of 4 items, which are family, friend, and a special person. In the Cronbach's Alpha Method that was used to measure the internal consistency, values were found to be between 0.80 and 0.95
Multidimensional Scale of Perceived Social Support (MSPSS) | 6-8 weeks postpartum
  The scale developed by Zimet et al. in 1988 and Turkish adaptation, validity and reliability studies were carried out by Eker, Arkar, and Yaldız (2001). The MSPSS is a 12-item scale, and includes 3 groups about the source of support, each of which consisting of 4 items, which are family, friend, and a special person. In the Cronbach's Alpha Method that was used to measure the internal consistency, values were found to be between 0.80 and 0.95
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | at 20 to 36 weeks gestational age
  The Turkish adaptation of the scale, developed in 2007 by Tennant et al., was done by Keldal in 2015. It is a five-point Likert-type scale, including 14 items. The lowest and the highest scores are 14 and 70 points. High scores indicate high mental wellbeing. Cronbach's alpha value of the scale was determined as 0.89
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | 6-8 weeks postpartum
  The Turkish adaptation of the scale, developed in 2007 by Tennant et al., was done by Keldal in 2015. It is a five-point Likert-type scale, including 14 items. The lowest and the highest scores are 14 and 70 points. High scores indicate high mental wellbeing. Cronbach's alpha value of the scale was determined as 0.89
The Wijma Delivery Expectancy/Experience Questionnaire B version (W-DEQ-B) | 6-8 weeks postpartum
  W-DEQ- B was developed by Wijma et al. to determine postpartum feelings and thoughts about the fear of women who gave vaginal birth (1998). The scale consists of a total of 33 6-point Likert-type questions. Each item is defined as 1 with a score between 1-6 and 6 as none. The minimum score on the scale is 33, while the maximum score is 198. The higher the scores, the higher the fear of birth experienced by women

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kaya, PhD, Principal Investigator — Zeynep Kamil Women and Children's Diseases Training and Research Hospital
Locations (3):
- Turkey (Türkiye) (3):
  - Saglık Bilimleri Universitesi, Istanbul
  - Zeynep Kamil Women's and Children's Diseases Training and Research Hospital, Istanbul
  - Kartal Dr.Lütfi Kırdar City Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No